CLINICAL TRIAL: NCT01386775
Title: Evaluation of Phenotypic and Genetic Properties in Male Subjects Affected By Hypohidrotic Ectodermal Dysplasia: Intrafamilial Variation
Brief Title: Male Subjects Affected By Hypohidrotic Ectodermal Dysplasia: Intrafamilial Variation
Status: Completed | Type: Observational
Sponsor: Edimer Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ECP-007
Record Dates: First submitted 2011-06-29; First posted 2011-07-01 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Hypohidrotic Ectodermal Dysplasia
Keywords: X-Linked Hypohidrotic Ectodermal Dysplasia; XLHED; Hypohidrotic Ectodermal Dysplasia; HED
MeSH Terms: conditions — Ectodermal Dysplasia 1, Anhidrotic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HED Affected Males
- Controls

SUMMARY:
This study in affected Hypohidrotic Ectodermal Dysplasia (HED) males and unaffected male controls, age 1 year and up, will use minimally invasive devices to image sweat ducts in intact skin, to measure stimulated sweat rate, and in a subset of subjects to collect clipped scalp hair samples for RNA analysis. This study is descriptive in nature and is intended to assess the ability to use innovative approaches to generate data from subjects over a wide age spectrum, with particular emphasis on phenotype variability between male siblings (same mutation).

DETAILED DESCRIPTION:
This pilot study in affected HED males and unaffected male controls, age 1 year and up, will use minimally invasive devices to image sweat ducts in intact skin, to measure stimulated sweat rate, and in a subset of subjects to collect clipped scalp hair samples for RNA analysis. This study is descriptive in nature and is intended to assess the ability to use innovative approaches to generate data from subjects over a wide age spectrum, with particular emphasis on phenotype variability between male siblings (same mutation). To this end, priority will be given to families that contain multiple affected siblings (i.e. two brothers). Summary data will be generated for the various groups tested, but no power calculations are involved.

ELIGIBILITY:
Inclusion Criteria:

* Registered and attending the 2011 NFED Family Conference;
* One year of age or greater;
* Conform to one of the following requirements for providing informed consent/assent:

  * if more than 18 years of age, subjects must provide signed informed consent;
  * if less than 18 years of age and it is determined that the subject is capable of providing assent, both the assent of the subject and consent of the parent(s) or guardian of that subject must be granted. Under this condition, both parents of the subject should give their permission, unless 1 parent is deceased, unknown, incompetent, or not available;
  * if the subject is incapable of providing assent, the consent of the parent(s) or guardian of the subject must be granted. Under this condition, both parents should give their consent, unless 1 parent is deceased, unknown, incompetent, or not available.
* As described in Section 3.2 above, subjects must meet one of the following criteria:

  * Male subjects with the clinical characteristics of HED, including at least a history of decreased sweating and either abnormal teeth (fewer permanent teeth, teeth are smaller than average and often have conical crowns), and/or sparseness of scalp and body hair (Male HED subjects with an affected sibling also enrolling in the study will be given priority to be in the study);
  * Healthy male controls, i.e. either unaffected male family members or unaffected male volunteers.

Exclusion Criteria:

* Known hypersensitivity to pilocarpine or pilocarpine-like muscarinic agonists;
* Known hypersensitivity to lidocaine or lidocaine like agents;
* Presence of pacemakers;
* Subjects who are not able or are not willing to comply with the procedures of this protocol;
* Subjects with any major medical problem that will prevent them from participating in this study.

Min Age: 1 Year | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Attendees of the National Foundation for Ectodermal Dysplasia's (NFED) 2011 Annual Family Conference
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Use skin assessment techniques to characterize skin properties in male subjects affected by HED compared with healthy controls, including determination of the number of sweat ducts and the rate of sweating | Day of study conduct
  Day 1

SECONDARY OUTCOMES:
Collecting demographic and clinical status information in male subjects affected by HED using a medical questionnaire | Day of study conduct
  Study Day 1
Assessment of intrafamilial phenotypic variability in families with multiple HED-affected male siblings | Day of study conduct
  Study Day 1 - Comparison of sweat duct counts, sweat rate and hair analysis among HED-affected male siblings
Evaluation of hair RNA profiles in samples from HED and unaffected male controls | Day of study conduct
  Study Day 1 -This is a novel use of the RNASeq technology and will follow the protocol provided by an expert in the field, Dr. Benjamin Yu. The hairs will be cut not plucked from the occipital scalp, with 10-20 collected hairs placed in a regular mailing envelope. The hair-containing envelopes will be shipped to Dr. Yu's laboratory for processing and analysis.
Confirming the presence of ectodysplasin A (EDA) gene mutations in HED subjects enrolled in this study | Day of study conduct
  Study Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy K Grange, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Hilton Garden Inn St. Louis Shiloh/O'Fallon, O'Fallon, Illinois, United States